CLINICAL TRIAL: NCT05689710
Title: The Action of Inositols and Alpha-lactalbumin on Glucose Metabolism, Arterial Stiffness and Vascular Damage in Patients With Metabolic Syndrome at Risk of Cardiac Fibrosis
Brief Title: The Effects of Inositol on Glucose Metabolism in Patients With Metabolic Syndrome at Risk of Cardiac Fibrosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in enrollment and patient compliance
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CARDIO_INO22
Record Dates: First submitted 2022-12-23; First posted 2023-01-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Syndrome; Cardiac Fibrosis
MeSH Terms: conditions — Metabolic Syndrome | interventions — Inositol; Lactalbumin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention)
- Experimental (Experimental): Dietary Supplement with inositols and alpha-lactalbumin
  Interventions: Dietary Supplement: Inositol and alpha-lactalbumin

INTERVENTIONS:
Dietary Supplement: Inositol and alpha-lactalbumin — The administration of an oral formulation based on inositol and alpha-lactalbumin (two sachets/day for 180 days)
  Arms: Experimental

SUMMARY:
The study aims to evaluate the effects of an oral supplementation based on inositols and alpha-lactalbumin on principals metabolic parameters in patients with metabolic syndrome at risk of cardiac fibrosis

ELIGIBILITY:
At least 3 of the following inclusion criteria:

* triglycerides levels ≥ 150 mg/dL
* HDL ≤ 40 mg/dL
* Fasting glycemia > 100 mg/dL <126 mg/dl
* Systolic Pressure ≥ 130 mmHg or Diastolic pressure ≥ 85 mmHg
* Hip circumference > 102 cm in men or 88 cm in women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | Four time points: changes in body weight (kg) from the baseline to 30, 90, 180 days

SECONDARY OUTCOMES:
Tryglicerides | Four time points: changes in blood levels of tryglycerides from the baseline to 30, 90, 180 days
  Plasmatic levels of tryglicerides
Hypertension | Four time points: changes in values of systolic and diastolic blood pressure from the baseline to 30, 90, 180 days
  sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Davide Grassi, MD, Principal Investigator — UOC Medicina Interna e Nefrologia P.O. AQ; Claudio Ferri, MD, Principal Investigator — UOC Medicina Interna e Nefrologia P.O. AQ
Locations (1):
- UOC Medicina Interna e Nefrologia P.O. AQ, L’Aquila, Italy